CLINICAL TRIAL: NCT04936750
Title: A One-arm, Prospective Study Comparing the Effects of Different Body Composition on the Survival of Patients Undergoing Radical Concurrent Chemoradiotherapy for Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LX202104022
Record Dates: First submitted 2021-06-16; First posted 2021-06-23 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2022-06

CONDITIONS: Brief Description of Focus of Study

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Analysis of body composition — The cross section of the third lumbar spine in the CT scan images of the patients was analyzed to obtain the parameters related to the body composition of the patients

SUMMARY:
Skeletal muscle depletion and sarcopenia are the most typical features of cachexia, which occurs in 80% of patients with advanced esophageal cancer. Skeletal muscle consumption is an independent factor for poor prognosis, which negatively affects therapeutic toxicity, length of hospital stay, quality of life, complications, infection, and survival. The vast majority of patients had already experienced severe weight loss and skeletal muscle loss before the treatment began. During the concurrent chemoradiotherapy period, the intensity and long cycle of treatment, the toxic and side effects of treatment and the occurrence of radiation esophagitis would further lead to the increased demand for energy and decreased intake of patients, thus leading to continuous weight loss. Based on the previous literature, we suggest that baseline body composition has a significant impact on nutritional status, the incidence of adverse reactions, and survival during treatment. This research mainly for the thorough chemoradiation in patients with esophageal cancer, analysis treatment precursor composition, including skeletal muscle index, visceral fat area, body fat percentage and other parameters on the side reaction of chemoradiation, nutritional status and the influence of survival, and observe the baseline body composition and cure after 1 month of body composition changes of the impact on the survival time.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and face to face signed informed consent;
* 18 -- 75 years old, gender unlimited;
* The histological diagnosis was esophageal squamous cell carcinoma, and the clinical staging was stage II-IVA (according to AJCC stage 8, pre-treatment clinical staging was: CT1N2-3M0, CT2-4BN0-3M0).
* Initial treatment patients receiving radical concurrent chemoradiotherapy; Immunotherapy with or without combination;
* The primary tumor can be evaluated;
* No distant metastasis;
* No serious abnormal function of blood system, heart, lung, liver and kidney or immune deficiency;
* Hemoglobin (Hb) ≥9 g/dL; White blood cell (WBC) ≥3×109/L; Neutrophils (ANC)≥1.5×109/L; Platelet (PT)≥100×109/L;
* Bilirubin < 1.5 times the upper limit of normal; Alanine aminotransferase (ALT) and alanine aminotransferase (AST) ≤2.5 times the upper limit of normal;
* Serum creatinine ≤1.5 times the upper limit of normal value;
* The willingness of men or women of reproductive age to use contraception in the trial;
* Physical condition score ECOG 0 ~ 2;
* The expected survival time was >3 months.

Exclusion Criteria:

* Patients who lacked an evaluation of CT body composition within 15 days prior to treatment initiation;
* Patients with severe intestinal function damage or inability to tolerate intestinal nutrition;
* The digestive tract is severely obstructed, unable to take food orally and unable/unwilling to undergo nasogastric tube or percutaneous gastrostomy;
* Previous surgery, chemoradiotherapy or bio-targeted therapy for esophageal cancer;
* Previous history of malignant tumor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal cancer receiving radical concurrent chemoradiotherapy with or without PD1 antibodies
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | one month
  To evaluate the effect of human components on the overall survival of patients with esophageal cancer undergoing radical concurrent chemoradiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital/, Tianjin, China